CLINICAL TRIAL: NCT00227812
Title: ERP-8654 - Integrated Treatment for Cocaine and Mood Disorders
Brief Title: Integrated Treatment for Cocaine and Mood Disorders - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Joy Schmitz, PhD, University of Texas Hlth Sci Ctr Houston
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08654-1; R01-DA08654-1; R01DA008654 (NIH)
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Cocaine Dependence; Depressive Disorder, Major
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Depressive Disorder, Major | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to test whether cognitive behavioral therapy and bupropion hydrochloride will help cocaine users, who are depressed, reduce or end their cocaine use and improve their mood.

DETAILED DESCRIPTION:
The global aim of this study is to evaluate an "integrated" treatment approach for cocaine dependent patients with comorbid unipolar depression. It is hypothesized that a cognitive-behavioral psychotherapy that targets both disorders, in combination with a pharmacotherapy, i.e., bupropion, is expected to provide the best coverage for dual disorders and thus maximize treatment outcomes. Specifically, we will conduct a double blind, placebo-controlled clinical trial involving the random assignment of participants into one of four treatment conditions according to a full 2x2 factorial research design. One independent variable will be pharmacotherapy (bupropion versus placebo); the other independent variable will be psychotherapy (integrated CBT versus clinical management). The study will enroll 140 cocaine dependent patients with comorbid major depressive disorder. A secondary objective is to further elucidate "primary" and "secondary" paradigms of depressive illness symptoms in cocaine-dependent adults and better understand how this distinction influences treatment outcome. This will be accomplished by enrolling a subsample of patients with substance-induced mood disorder. Taken together, this proposal will examine the feasibility and relative efficacy of a novel integrated treatment model for dually-diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* Generally physically healthy
* Aged 18-55
* Meets cocaine dependence by DSM-IV criteria
* Meets major depressive disorder or substance-induced depression disorder by DSM-IV criteria.
* Willing and able to participate in the 12 week treatment study and one year follow up.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Taking medications that interact with the study medication (MAO inhibitors, anticonvulsants, haloperidol, phenothiazines,selegiline, anesthetics
* Have other psychiatric diagnoses requiring therapy or medication.
* Physically dependent on opiates or alcohol.
* Currently being treated with bupropion hydrochloride (e.g. Zyban).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 2001-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Urine toxicology for cocaine

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schmitz, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Sci Cntr Houston, Houston, Texas, United States